CLINICAL TRIAL: NCT00637390
Title: A Phase I Study of Alemtuzumab in Patients With Relapsed Ovarian/Primary Peritoneal Cancer.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Genzyme will no longer supply the study drug for this trial as it does not believe the study will not fully enroll within an appropriate time frame.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.120
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one (Experimental)
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — will be given Alemtuzumab therapy three times in your first week on the study and then once a week for six additional weeks

SUMMARY:
Ovarian cancer cannot grow without recruiting new blood vessels. Studies in humans have identified a novel cell population, termed vascular leukocytes (VLCs). While VLCs are not cancer cells, they support the growth of ovarian cancer cells by stimulating the growth of new blood vessels which provide the cancer with nutrients. VLCs make a protein termed CD52. An antibody therapeutic, Alemtuzumab (also know as Campath), that kills cells that make the CD52 protein has been successfully used to treat certain lymphomas (a type of blood cell cancer) that make CD52 protein. The purpose of this study is to determine if Alemtuzumab given subcutaneously (under the skin)can be safely given to patients with ovarian, fallopian, or primary peritoneal cancers to kill VLCs and determine if Alemtuzumab, by eliminating VLCs, can restrict tumor growth or increase response rates to chemotherapy given after the discontinuation of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of histologically confirmed ovarian, fallopian or primary peritoneal cancer that has progressed or recurred in the abdomen or pelvis after salvage chemotherapy as documented by either:

   1. Radiologic studies or
   2. Rising CA125 levels on two independent measurements. If the patient's CA125 has fallen into a normal range, CA125 relapse will be defined as double the nadir CA125. However, if the patients CA125 nadir had fallen to less than 10, then the measurements documenting recurrence or progression must be greater than 20.
2. There is no limit on prior courses of chemotherapy.
3. Patients must have unidimensional measurable disease or elevated CA125
4. Age greater than 18 years.
5. ECOG performance status less tha 2 (Karnofsky 60%).
6. Life expectancy of greater than 12 weeks.
7. Patients must have adequate organ and marrow function
8. Ability to understand and the willingness to sign a written informed consent document. All patients must be informed of the investigational nature of this study and must sign an informed consent in accordance with institutional and federal guidelines.
9. Timing guideline for pre-study labs and measurements:

All pre-study labs required for determination of eligibility are to be completed within 28 days of treatment Day 1.

X-rays and/or scans used for tumor measurement to determine disease status are to be completed within 28 days of treatment Day 1.

Women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Patients with known immunosuppressive diseases are excluded from this trial due to the known immunosuppressive nature of Alemtuzumab therapy.
2. Patients may not be receiving any other agents (investigational or otherwise) with therapeutic intent.
3. Patients with prior malignancy, except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease free for 2 years.
4. Patients with a history of allergic reactions to Alemtuzumab or other humanized immunotherapeutics.
5. Patients with unresolved bacterial, fungal, or viral infections requiring active treatment. Patients may be registered two weeks after the conclusion of antibiotic or anti-viral therapy.
6. Patients with history of active CMV disease as Alemtuzumab therapy has been associated with CMV reactivation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
safety & maximally tolerated dose | Maybe 2 years

SECONDARY OUTCOMES:
Effectiveness of Alemtuzumab to eliminate VLCs. | Maybe 2 years
Assess molecular markers associated with reduction in VLCs. | Maybe 2 years
Anti-tumor activity measured by decline or stabilization of CA125(a protein that is a tumor marker)or radiological(ie. CT, MRI, X-Ray)improvement or improvement in progression free survival. | Maybe 2 years
Alemtuzumab effect on patients' response rates to chemotherapy given after the discontinuation of chemotherapy. | Maybe 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States